CLINICAL TRIAL: NCT05162703
Title: Evaluation of Exercise Induced Bronchoconstriction by Field Test Using Lung Function and a Novel Automated Digital Clinical Decision System (DFET)
Brief Title: Evaluation of Exercise Induced Bronchoconstriction Using a Novel Automated Digital Clinical Decision System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: K 2021-5960
Record Dates: First submitted 2021-11-12; First posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-11

CONDITIONS: Exercise Induced Asthma; Exercise Induced Bronchospasm; Pediatric Respiratory Diseases
MeSH Terms: conditions — Asthma, Exercise-Induced

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Participants will be equipped with a spirometer and and the AsthmaTuner mobile phone app to perform an exercise tests in their natural training environment. Feasibility will be evaluated using questionnaires.
  Interventions: Diagnostic Test: AsthmaTuner

INTERVENTIONS:
Diagnostic Test: AsthmaTuner — Exercise challenge test using AsthmaTuner mobile phone app and spirometer.

SUMMARY:
The primary objective of this study is to assess if the unstandardized field exercise challenge test (ECT) using AsthmaTuner can be performed independently by youths that have been investigated for asthma. This is an open feasibility study including youths who have been investigated for asthma. Participants will be equipped with a digital spirometer and mobile phone app to perform an exercise tests in their natural training environment. Feasibility will be evaluated using questionnaires.

DETAILED DESCRIPTION:
Asthma is the most common chronic condition in athletes and people who exercise regularly. Asthma is defined as a chronic inflammation in the airways associated with bronchial hyper responsiveness (BHR). While exercise-induced "sports" asthma (EIA) describes symptoms and signs of asthma provoked by exercise, exercise-induced bronchoconstriction (EIB) is defined as the transient narrowing of the lower airway after exercise. In the general population, EIB with or without asthma affects 5% to 20%, but the rate is estimated to be even higher in top athletes participating in winter and summer endurance sports.

Asthma and EIB represents an important challenge in both athletes and the general population, and correct diagnosis is important as it affects health as well as performance.

Presence of BHR is demonstrated by direct or indirect bronchial provocation testing. Indirect bronchial provocation includes several methods for the diagnosis of EIB. The most intuitive is exercise (field and laboratory) challenge testing (ECT), but sensitivity has been reported to be low, since exercise load and intensity have large impact on ability to detect EIB and in field-testing (FT), standardizing ambient conditions are impossible.

Suboptimal tests for EIB may explain why previous papers report poor relationship between symptoms of EIA and the objective EIB in athletes, leaving the actual rate of EIB remains unclear. What has been argued to be the true "gold standard" is a sports-specific exercise FT, performed in the actual training conditions which also makes it easier for the athlete to perform at maximum exercise. The advantages of monitoring with peak expiratory flow (PEF) or forced expiratory volume in 1 s (FEV1) outside a laboratory with a PEF meter or spirometer, respectively, are that it is simple and cheap. It also enables measure of bronchial challenge testing in close relationship to symptoms, since laboratory bronchial challenge testing often are negative in subjects being away from their profession too long. However, traditional non-digital method of serial PEF/FEV1 monitoring has limitations with poor adherence, interpretation difficulties with objectivity and time-consuming analysis and reading of paper PEF/FEV1 plots.

Recently, AsthmaTuner (Medituner AB) consisting of a patient smartphone application, a portable wireless spirometer for measuring lung function (PEF/FEV1), and a healthcare interface including treatment plan, was reported to significantly improve management of uncontrolled asthma. Such electronically clinical decision support systems (CDSS) has gained acceptance for the diagnosis of asthma, and by the ability to assess patient generated data in field ECTs, the CE-marked AsthmaTuner may provide athletes a feasible, time and cost-efficient self-monitoring of EIB and asthma. AsthmaTuner may also empower athletes in monitoring their lung function over time. These lung function measurements contain unexpected amounts of information for identifying athletes with distinct phenotypes of EIB due to strenuous sports and environmental conditions. Hence, AsthmaTuner have the potential to fill the knowledge gap regarding prevalence of EIB, development of EIB and the lack of association between symptoms and detection of EIB in athletes.

The primary objective of this study is to assess if the unstandardized field exercise challenge test (ECT) using AsthmaTuner can be performed independently by youths that have been investigated for asthma. This is an open feasibility study including youths who have been investigated for asthma. Participants will be equipped with a spirometer and and the AsthmaTuner mobile phone app to perform an exercise tests in their natural training environment. Feasibility will be evaluated using questionnaires.

ELIGIBILITY:
Inclusion criteria:

Current or previous investigation for exercise induced asthma and have performed a standardised exercise challenge test at Astrid Lindgren's Children's Hospital in the last 2 years.

Exclusion Criteria:

Other medical conditions or medications that interfere with asthma or respiratory tract infection in the last two weeks.

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-03-14 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Ability to perform test | 2 weeks
  Number of participants who completed the test

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Ljungberg, Study Chair — henrik.ljungberg@regionstockholm.se
Locations (1):
- Astrid Lindgren Children's Hospital, Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No